CLINICAL TRIAL: NCT02569346
Title: Bioequivalence Study of CRushed TriUMeq With or Without Drip Feed Compared to the Whole Tablet (SCRUM)
Brief Title: Bioequivalence Study of CRushed TriUMeq With or Without Drip Feed Compared to the Whole Tablet
Acronym: SCRUM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 15.02
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: HIV
Keywords: Triumeq; Pharmacokinetics; Crushing; Drip feed
MeSH Terms: conditions — Pressure Ulcer | interventions — abacavir, dolutegravir, and lamivudine drug combination; Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triumeq whole (Active Comparator): Single-dose Triumeq as a whole tablet in a fasted state
  Interventions: Drug: Triumeq crushed + breakfast; Drug: Triumeq crushed + drip feed
- Triumeq crushed + breakfast (Experimental): Single-dose crushed and suspended Triumeq in a fasted state
  Interventions: Drug: Triumeq; Drug: Triumeq crushed + drip feed
- Triumeq crushed + drip feed (Experimental): 250 ml drip feed (Nutrison) followed by a single-dose crushed and suspended Triumeq
  Interventions: Drug: Triumeq; Drug: Triumeq crushed + breakfast

INTERVENTIONS:
Drug: Triumeq — Single-dose Triumeq as a whole tablet
  Arms: Triumeq crushed + breakfast; Triumeq crushed + drip feed
Drug: Triumeq crushed + breakfast — Single-dose crushed and suspended tablet of Triumeq
  Arms: Triumeq crushed + drip feed; Triumeq whole
Drug: Triumeq crushed + drip feed — Drip feed followed by single-dose crushed and suspended tablet of Triumeq
  Arms: Triumeq crushed + breakfast; Triumeq whole

SUMMARY:
Dolutegravir is an HIV-1 integrase inhibitor which is marketed as a single tablet (Tivicay®) and in a fixed dose combination tablet with abacavir and lamivudine (Triumeq®, referred to as TRI). For patients with swallowing difficulties, administration of whole tablets can be problematic and tablets are cut or crushed to ease administration.

Currently there is no information about crushing TRI tablets. Therefore this study will be conducted to investigate whether crushed and suspended TRI and crushed and suspended TRI with drip feed are bioequivalent to taking TRI as a whole.

DETAILED DESCRIPTION:
Dolutegravir is an HIV-1 integrase inhibitor which is marketed as a single tablet (Tivicay®) and in a fixed dose combination tablet with abacavir and lamivudine (Triumeq®, referred to as TRI). For patients with swallowing difficulties, administration of whole tablets can be problematic and tablets are cut or crushed to ease administration. In addition, if HIV patients develop opportunistic infections, patients can become severely ill and may end up on the intensive care. Patients at the intensive care might not be able to swallow medication. Therefore it is useful to know if it is possible to administer TRI through a different route, like a feeding tube. If TRI can be crushed or dissolved and given through a catheter it is also useful to know if it can be given with drip feed.

Currently there is no information about crushing TRI tablets. Depending on the biopharmaceutical characteristics of a drug formulation, crushing tablets can lead to altered pharmacokinetics of drugs. This has been shown for some of the antiretroviral drugs, such as ritonavir, lopinavir, efavirenz and tenofovir.

It is important to know whether pharmacokinetics are influenced by crushing of tablets as low concentrations are associated with virologic failure. Therefore higher doses or switching to other HIV-drugs might be needed. In addition, higher Cmax and/or exposure can lead to toxicity. As a result therapeutic drug monitoring is advised, or crushing the drug is a contra-indication based on the available data.

It has been shown that DTG plasma concentration is influenced by food, with higher AUC en Cmax after a high-fat meal compared to administration in a fasted state. During clinical development, however, dolutegravir intake was studied without regard to food intake. Therefore, it is recommended that dolutegravir can be taken with or without food.

In addition, it has been shown that simultaneous oral ingestion of antacids and dolutegravir gives a decrease in Cmax and AUC of dolutegravir. This interaction is not shown for co-ingestion with omeprazole, which makes it unlikely that this interaction is caused by a pH-lowering effect influencing the absorption of dolutegravir. It is probably a local gastrointestinal complexation phenomenon, similar to what has been observed with other HIV integrase inhibitors. A possible pharmacokinetic interaction between dolutegravir and complexation formers may be expected. Especially considering the active binding sites of dolutegravir which bind magnesium metal ion cofactors. It is currently unclear if certain foods or liquids containing high amounts of magnesium or other cations, like drip feed, can cause this same interaction.

Therefore this study will be conducted to investigate whether crushed and suspended TRI and crushed and suspended TRI with drip feed are bioequivalent to taking TRI as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years of age at the day of screening.
* Subject weighs at least 40 kg.
* Subject has a BMI of 18.5-30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within four weeks prior to day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included based on the Investigator's judgment that the observed deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgment.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to day 1.

Exclusion Criteria:

* Positive HIV test.
* Positive hepatitis B or C test.
* Positive HLA-B*5701 status (the risk for abacavir hypersensitivity reaction to occur is high for subjects who test positive for the HLA-B*5701 allele).
* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the study and the procedures required.
* Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
* Therapy with any drug (including herbal remedies, multivitamins, magnesium- and calcium-containing supplements, etc.) (for two weeks preceding day 1), except for acetaminophen.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal disorders (renal failure determined as an estimated Glomerular Filtration Rate (eGFR) below 50 ml/min (MDRD-based)), hepatic disorders (Child-Pugh B or C), hormonal disorders (especially diabetes mellitus), coagulation disorders.
* History of or current abuse of drugs, alcohol or solvents.
* Gluten free diet.
* Participation in a drug study within 60 days prior to day 1.
* Donation of blood within 60 days prior to day 1.
* Febrile illness within 3 days before day 1.
* Co-worker of Radboud university medical center.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AUC | up to 48 hours after administration

SECONDARY OUTCOMES:
Adverse events | during the entire conduct of the study, 6 weeks in total

CONTACTS AND LOCATIONS:
Locations (1):
- CRCN, Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Roskam-Kwint M, Bollen P, Colbers A, Duisenberg-van Essenberg M, Harbers V, Burger D. Crushing of dolutegravir fixed-dose combination tablets increases dolutegravir exposure. J Antimicrob Chemother. 2018 Sep 1;73(9):2430-2434. doi: 10.1093/jac/dky191. PMID 29796595